CLINICAL TRIAL: NCT00719290
Title: A Randomised Comparative Study of the Effects of Cataract Extraction With Lens Implant Alone Versus Cataract Extraction With Lens Implant and Goniosynechialysis on Outflow Facility in Patients With Primary Angle Closure Glaucoma.
Brief Title: Primary Angle Closure Glaucoma and Aqueous Dynamics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, KIN SHENG LIM, Consultant Ophthalmic Surgeon, Guy's and St Thomas' NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RJ1 08/0124
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Primary Angle Closure
Keywords: Primary Angle Closure Glaucoma; Phacoemulsification; Goniosynechialysis; Outflow facility
MeSH Terms: conditions — Glaucoma, Angle-Closure | interventions — Phacoemulsification; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Phacoemulsification with intraocular lens implant alone
  Interventions: Procedure: Phacoemulsification (Acrylic Foldable Intraocular Lens (Acrysoft)), (Healon5)
- 2 (Active Comparator): Phacoemulsification with intraocular lens implant and goniosynechialysis
  Interventions: Procedure: Phacoemulsification and goniosynechialysis (Acrylic Foldable Intraocular Lens (Acrysoft)), (Healon5)

INTERVENTIONS:
Procedure: Phacoemulsification (Acrylic Foldable Intraocular Lens (Acrysoft)), (Healon5) — Phacoemulsification of the lens with intraocular lens implant
  Other Names: Healon5; Acrylic Foldable Intraocular Lens (Acrysoft)
  Arms: 1
Procedure: Phacoemulsification and goniosynechialysis (Acrylic Foldable Intraocular Lens (Acrysoft)), (Healon5) — Phacoemulsification of the lens with intraocular lens implant and goniosynechialysis
  Other Names: Healon5; Acrylic Foldable Intraocular Lens (Acrysoft)
  Arms: 2

SUMMARY:
The aim of the study is to determine which is the best treatment for people with cataract and primary angle closure (PAC).In PAC, apposition of the iris tissue to the drainage channels (Trabecular Meshwork-TM) of the eye results in damage and formation of adherences between these structures (Peripheral anterior synaechiae-PAS) causing a mechanical obstruction of the aqueous outflow via the TM. It is thought that cataract surgery combined with mechanical separation of the iris from the TM with the breakage of PAS(we call this separation 'goniosynechialysis') would make the pressure even lower as it would cause the drain to open to a greater extent than cataract surgery alone. This technique is not new, and the results have been very encouraging. Comparing this technique to cataract surgery alone however, has not been done and this is exactly what we would like to do in order to help us decide what is the best treatment.

In summary, the investigators propose that cataract surgery with goniosynechialysis would lower intraocular pressure to a greater extent than cataract surgery alone in patients with significant PAS.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years.
* Diagnosis of PAC or PACG. PACG is defined as glaucomatous optic neuropathy in the opinion of a fellowship-trained glaucoma specialist, together with an IOP > 21mmHg on at least one occasion, and reproducible visual field defect (using the 24-2 test pattern on a Humphrey Field Analyser). PAC has all the above characteristics except for the visual field defect.
* More than 90 degrees of PAS (not necessarily contiguous).
* Lens opacity deemed sufficient to be causing decreased vision in the opinion of the supervising consultant (KSL).
* Ability to give informed consent.

Exclusion Criteria:

* Previous intraocular surgery or keratorefractive surgery.
* Previous eye trauma resulting in documented damage to the drainage angle (such as angle recession).
* History of uveitis.
* For patients on warfarin, INR >3.0 on day of surgery.
* Anterior segment neovascularisation.
* Chronic use of topical or systemic steroids.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-07; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
1. Outflow facility Success defined as increased outflow facility at 3 month compared to baseline with the same or reduced number of intraocular pressure lowering medications. | 3 months

SECONDARY OUTCOMES:
1. Intraocular pressure Success defined as decreased IOP at 3 month compared to baseline with the same or reduced number of intraocular pressure lowering medications | 3 months
Intra- or post operative complications | 2-3 weeks
Long-term PAS development | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: K Sheng Lim, MB ChB MD FRCOpht, Principal Investigator — Guys ans St Thomas' NHS Trust
Locations (1):
- St Thomas' Hospital, London, United Kingdom

REFERENCES:
- [Derived] Rodrigues IA, Alaghband P, Beltran Agullo L, Galvis E, Jones S, Husain R, Lim KS. Aqueous outflow facility after phacoemulsification with or without goniosynechialysis in primary angle closure: a randomised controlled study. Br J Ophthalmol. 2017 Jul;101(7):879-885. doi: 10.1136/bjophthalmol-2016-309556. Epub 2016 Oct 17. PMID 28400374